CLINICAL TRIAL: NCT07149545
Title: Electrophysiologist-led Deep Sedation Protocols for Pulsed Field Ablation for Atrial Fibrillation Using a Bipolar Tip-Catheter: The DEEP-PFA Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS2025277
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation (AF); PFA; Deep Sedation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fentanyl; Midazolam; flurbiprofen axetil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Fentanyl + Midazolam) (Experimental): After venipuncture, patients receive intravenous midazolam 0.5 mg and fentanyl 20 µg, followed by continuous fentanyl infusion at 1-1.5 µg/kg/h. An additional 0.5 mg of midazolam is administered before interatrial septal puncture. After the start of ablation, fentanyl infusion is increased to 2.0-2.5 µg/kg/h. If needed, 0.5 mg of midazolam or 2 mL of fentanyl may be added.
  Interventions: Drug: Arm A (Fentanyl + Midazolam)
- Arm B (Flurbiprofen axetil + Fentanyl + Midazolam) (Experimental): After venipuncture, patients receive midazolam 0.5 mg and fentanyl 20 µg intravenously, followed by a fentanyl infusion at 1-1.5 µg/kg/h. Prior to septal puncture, patients receive flurbiprofen axetil 50-100 mg and an additional 0.5 mg of midazolam. After ablation begins, fentanyl infusion is increased to 2.0-2.5 µg/kg/h. If needed, 0.5 mg of midazolam or 2 mL of fentanyl may be added.
  Interventions: Drug: Arm B (Flurbiprofen axetil + Fentanyl + Midazolam)
- Arm C (Fentanyl + Dexmedetomidine) (Experimental): Following femoral venous access, a loading dose of dexmedetomidine (1.0 µg/kg) was infused intravenously over 15 minutes. A maintenance infusion of 0.4 µg/kg/h was initiated thereafter (typically post-transseptal puncture). Fentanyl infusion commenced at venous access (1.0-1.5 µg/kg/h) and was increased to 2.0-2.5 µg/kg/h during ablation. Rescue boluses of midazolam (0.5 mg) or fentanyl (20-50 µg) were administered if required.
  Interventions: Drug: Arm C (Fentanyl + Dexmedetomidine)

INTERVENTIONS:
Drug: Arm A (Fentanyl + Midazolam) — Prior to venous puncture, administer 0.5 mg midazolam intravenously, concurrently with 20 µg fentanyl intravenously. Subsequently, maintain fentanyl infusion at 1-1.5 µg/kg/h. Prior to atrial septal puncture, administer an additional 0.5 mg midazolam. Upon initiation of ablation, adjust the fentanyl infusion rate to 2.0-2.5 µg/kg/h. If required during ablation, supplement with 0.5 mg midazolam or 2 ml fentanyl.
  Arms: Arm A (Fentanyl + Midazolam)
Drug: Arm B (Flurbiprofen axetil + Fentanyl + Midazolam) — Prior to venous puncture, administer 0.5 mg midazolam intravenously, followed by 20 µg fentanyl intravenously. Subsequently, maintain fentanyl infusion at 1-1.5 µg/kg/h. Prior to atrial septal puncture, administer 50-100 mg flurbiprofen ester and 0.5 mg midazolam. Upon ablation initiation, adjust the fentanyl infusion rate to 2.0-2.5 µg/kg/h. If required during ablation, supplement with 0.5 mg midazolam or 2 ml fentanyl.
  Arms: Arm B (Flurbiprofen axetil + Fentanyl + Midazolam)
Drug: Arm C (Fentanyl + Dexmedetomidine) — Prior to venous puncture, administer dexmedetomidine intravenously at 1 µg/kg/h for 15 minutes, then reduce to 0.4 µg/kg/h. Concurrently, administer fentanyl intravenously at 20 µg. Subsequently, maintain dexmedetomidine infusion at 1-1.5 µg/kg/h. After ablation initiation, adjust the fentanyl infusion rate to 2.0-2.5 µg/kg/h. If required during ablation, administer an additional 0.5 mg midazolam or 2 ml fentanyl.
  Arms: Arm C (Fentanyl + Dexmedetomidine)

SUMMARY:
The DEEP-PFA trial is an investigator-initiated, prospective, single-center, three-arm (1: 1: 1), randomized controlled study comparing three anesthesia regimens-midazolam + fentanyl (DS1), flurbiprofen + midazolam + fentanyl (DS2), and dexmedetomidine + midazolam + fentanyl (DS3)-for non-airway-assisted pulsed-field ablation (PFA) in atrial fibrillation (AF). Patients scheduled for atrial fibrillation ablation at Beijing Anzhen Hospital will be screened for eligibility. Following signature of informed consent, patients who meets all inclusion criteria without any exclusion criteria, will be randomly assigned at a 1:1:1 ratio to one of three groups: (1) DS1: Traditional Midazolam Group (Midazolam + Fentanyl); (2) DS2: Enhanced Analgesia Group (Flurbiprofen + Midazolam + Fentanyl); or (3) DS3: Enhanced Sedation Group (Dexmedetomidine + Midazolam + Fentanyl). The primary endpoint of this study was the proportion of patients achieving a Ramsay sedation score of ≥3 at the start of ablation.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-80 years
2. Diagnosis of paroxysmal or persistent atrial fibrillation with clinical indication for catheter ablation
3. Planned use of PFA as the ablation strategy
4. Ability and willingness to provide written informed consent

Exclusion criteria:

1. Known hypersensitivity or allergy to study medications (fentanyl, midazolam, dexmedetomidine, flurbiprofen axetil)
2. Heart failure NYHA class III-IV
3. Severe obstructive sleep apnea syndrome
4. Severe respiratory disease, significant hepatic or renal dysfunction, advanced malignancy, or comorbidities with expected survival <1 year
5. Pregnancy or breastfeeding
6. Refusal to participate
7. Other circumstances deemed unsuitable for participation by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-01-27 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with successful sedation at the start of ablation | At the initiation of ablation
  The primary endpoint of this study was the proportion of patients achieving a Ramsay sedation score of ≥3 at the initiation of ablation. The Ramsay sedation scale is as follows: 1 indicates restlessness; 2 indicates fully awake, quiet, and cooperative; 3 indicates drowsy but responsive to verbal commands; 4 indicates lightly asleep but responsive to touch or pain; 5 indicates asleep but slowly responsive to touch or pain; and 6 indicates deeply asleep with no response.

SECONDARY OUTCOMES:
Incidence of hypotension | Perioperative period
  Defined as a mean arterial pressure (MAP) <65 mmHg or a ≥20% reduction from baseline.
Incidence of hypoxemia | perioperative period
  Defined as SpO₂ <90% lasting for over 10 s.
Number of intraoperative interventions | perioperative period
  Number of intraoperative interventions (oxygen adjustment, hemodynamic drugs, airway management, conversion to general anesthesia)
Sedation difficulty score. Score on a 5-point Likert scale (1=Very dissatisfied, 5=Very satisfied). | Perioperative period
  Rated by the operating electrophysiologist on a 5-point Likert scale (1 = not difficult, 2 = mildly difficult, 3 = moderately difficult, 4 = very difficult, 5 = extremely difficult).
Operator satisfaction. Score on a 5-point Likert scale (1=Very dissatisfied, 5=Very satisfied). | perioperative period
  Operator satisfaction (5-point Likert scale): Rated postoperatively by the operating electrophysiologist on a 5-point Likert scale (1 = very dissatisfied, 2 = somewhat dissatisfied, 3 = neutral, 4 = satisfied, 5 = very satisfied).
Patient recall of intraoperative pain. Score on a 10-point Visual Analog Scale (0=No pain, 10=Worst pain). | perioperative period
  Intraoperative pain intensity: Measured postoperatively based on patient recall using a 10-point Visual Analogue Scale (VAS, 0 = no pain, 10 = worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No